CLINICAL TRIAL: NCT00169754
Title: Do Calcium Oxalate Renal Calculi Originate From Randall's Plaque?
Brief Title: Attached Stone Project: Do Calcium Oxalate Renal Calculi Originate From Randall's Plaque?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Dr. James E. Lingeman, Methodist Urology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-031
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Renal Calculi
Keywords: Nephrolithiasis; Renal Calculi; Perc; Attached Stones
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cohort (Other): mapping and data collection
  Interventions: Other: mapping kidney anatomy

INTERVENTIONS:
Other: mapping kidney anatomy — videotape of surgical procedure to document location of attached stones and condition of calyces and papilla.

SUMMARY:
Urolithiasis is a common condition in the United States, and is associated with significant morbidity and even mortality. The most commonly occurring urinary calculi are comprised of calcium oxalate salts, and until recently, the pathogenesis of calcium oxalate calculi was poorly understood. New evidence, however, suggests that the development of calcium oxalate calculi may be intimately associated with hydroxyapatite (HA) plaque, also known as Randall's plaque, which is located on the renal papillae. The investigators have previously demonstrated that Randall's plaque originates in the thin ascending limb of the loop of Henle, and they have shown that Randall's plaque is composed of HA (Evan, Lingeman et al. 2003). As well, the amount of Randall's plaque correlates with elevated levels of urinary calcium and decreased urinary volume, risk factors for the formation of calcium oxalate calculi (Kuo, Lingeman et al. 2003). In the course of these previous studies, the investigators have anecdotally noted that calcium oxalate stones are often found attached to Randall's plaque, an observation that others have reported as well (Prien 1949; Carr 1954; Cifuentes Delatte, Minon-Cifuentes et al. 1987). However, there has been no in-vivo, rigorous documentation of this "attached stone" relationship. Attached calculi represent an important point in the pathogenesis of calcium oxalate calculi, as they correspond to a moment in time where there is a continuum between the HA plaque of Randall and the calcium oxalate stone, thus linking the origin of plaque with the development of stone. A better understanding of the phenomenon of attached calculi will lead to a better understanding of how and why calcium oxalate stones form, which may ultimately direct future interventions to attenuate stone activity.

DETAILED DESCRIPTION:
Urolithiasis is a very common condition in the United States, with an estimated prevalence of 11.7% by age 70. Furthermore, it has been associated with considerable patient morbidity and occasional mortality (Stamatelou, Francis et al. 2003). Direct costs associated with the treatment of renal calculi are enormous, as over 600,000 stone related medical procedures are performed annually in the United States (shock wave lithotripsy (SWL), ureteroscopy (URS), percutaneous nephrolithotomy (PERC), stone removal, ureteral stents, and stone basketing (source: Boston Scientific Corporation). Although the last two decades have seen considerable advances in less invasive techniques for the treatment of symptomatic stone episodes, as well as progress in mitigating the risks of new stone formation, our knowledge of the inciting lesion in human urolithiasis remains rudimentary and much debated.

Until recently, the sequence of events that leads to the formation of urinary calculi were poorly understood, most fundamentally due to the lack of appropriate in-vivo data. Earlier theories of calculogenesis proposed that stones could result from tubular epithelial injury due to oxalate toxicity, a lack of urinary inhibitors of crystal formation or crystal epitaxy on a pre-existing nidus (Khan, Finlayson et al. 1979). Theoretical work on free and fixed particle growth indicated that a transit time from the collecting duct to the bladder of only 10 minutes provided insufficient time for a crystal to grow to a clinically meaningful size (Jonassen, Cooney et al. 1999). Morphological classification of the directional growth of calculi supported the necessity for a fixed point of origin, in the absence of obstruction (Hinman 1979). These observations suggested that most stones must initiate from a fixed point or nidus in the collecting system or renal papilla.

One such nidus, first described more than sixty years ago by Alexander Randall, was proposed to be the originating lesion for the formation of calcium oxalate stones (Randall 1936; Randall 1937; Randall 1940). In microscopic studies of renal papilla obtained at necropsy, he demonstrated the presence of 2-3mm lesions in 19.6% of patients that were composed of calcium phosphate and devoid of evidence of inflammation. Adherent to this, in 65 of 1,514 pairs of kidneys, he identified nascent stones composed of calcium oxalate and calcium phosphate. When these stones reached sufficient size, he hypothesized that they would break free, taking with them the underlying plaque. In subsequent work, 256 voided or removed calculi were examined and 106 gave visible evidence of mural attachment (Randall 1940). Later microradiographic studies would confirm the presence of plaque in a papillary location that could be co-localized with stone (Carr 1954). Unfortunately, all earlier studies of stone pathogenesis have suffered from lack of definition of clear clinical stone-forming phenotypes.

There are intriguing reports to support Randall's, and our, hypothesis that stones originate from a fixed plaque composed of HA. Earlier microscopic studies of stone structure demonstrated the presence of concavities on small stones compatible with a point of mural attachment and indicated that apatite may be present at the attachment point (Rosenow 1940; Prien 1949). In an early x-ray diffraction and crystallographic study of 10,000 urinary calculi, Herring noted that HA was frequently found as the nucleus of calcium oxalate monohydrate, usually as a small discoid plaque which was felt to resemble Randall's plaque (Herring 1962). Later, Chambers performed an electron probe analysis of 115 small renal calculi. Of 92 predominantly calcium oxalate stones, he was able to identify small central areas of HA, usually 10-200 microns in diameter, in 70 (Chambers, Hodgkinson et al. 1972). Using scanning electron microscopy and x-ray dispersive energy, Cifuentes Delatte found that 63 of 87 passed calcium oxalate stones had evidence of plaque (Cifuentes Delatte, Minon-Cifuentes et al. 1985). Observation of uncalcified tubular lumens found in conjunction with these plaques suggested an interstitial papillary tip origin of this material (Cifuentes Delatte, Minon-Cifuentes et al. 1987).

We have noted that when endoscopically examining the renal papillae of patients undergoing PERC, oftentimes stones attached to renal papillae are encountered. We have collected three attached stones from three separate patients who were undergoing PERC. The stones were analyzed with a Micro CT device, and 3-D reconstruction with identification of mineral components was performed. The stones all showed multiple mineral components, including calcium oxalate, apatite, and probable regions of poorly mineralized matrix. Although the significance of these various components, in varying amounts, is not yet well understood, it is apparent that even at early stages of stone formation, multiple minerals in complex arrangement are present in papilla-attached stones. It will be only through a rigorous, prospectively designed protocol that the significance of attached renal calculi will be understood. By demonstrating that renal calculi in a population of common calcium oxalate stone formers originate from an HA plaque, we would link in a substantive way the origin of plaque with the subsequent development of stone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of Methodist Urology in Indianapolis, IN with kidney stones appropriate for percutaneous lithotripsy (PERC)
* Age greater than 18 years

Exclusion Criteria:

* Inability to give informed consent
* Active infection
* Bleeding diathesis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Detailed analysis of all stones from common calcium oxalate stone formers to determine stone composition and the site of stone attachment | one year

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — Methodist Urology, LLC
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States